CLINICAL TRIAL: NCT01044186
Title: A Protocol to Allow Treatment With ICL670 for Patients With or at Risk of Life-threatening Complications of Transfusional Iron Overload Who Are Unable to Tolerate Other Iron Chelators Because of Documented Severe Toxicity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICL670A0117; 2004-002303-32 EudraCT number (Registry Identifier: 2004-002303-32)
Record Dates: First submitted 2010-01-05; First posted 2010-01-07 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Transfusional Iron Overload
Keywords: Deferasirox; ICL670A; Iron chelators; Deferiprone; Transfusional hemosiderosis; Congenital aplastic anemia (Diamond Blackfan anemia); Red cell aplasia; Thalassemia; β thalassemia
MeSH Terms: conditions — Cystinosis; Anemia, Diamond-Blackfan; Red-Cell Aplasia, Pure; Thalassemia | interventions — Deferasirox

ARMS (1):
- ICL670 (Experimental)
  Interventions: Drug: ICL670

INTERVENTIONS:
Drug: ICL670

SUMMARY:
The purpose of this open-label, non-comparative, multi-center protocol was to further evaluate safety and to provide treatment with ICL670 to patients who had or were at risk of life threatening complications due to transfusional iron overload with a documented inability to tolerate any of the commercially available iron chelators due to severe toxicity rendering continued therapy either impossible or hazardous. Patients who were also ineligible for all on-going registration trials with ICL670 were included in the study. In exceptional cases, patients with a degree of iron overload which was not immediately life-threatening and who were ineligible for the registration trials were also enrolled provided they had a well-documented, sound justification for alternative chelation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients had to be at risk of life-threatening complications due to transfusional iron overload and be unable to tolerate therapy with any of the commercially available iron chelators (mainly deferoxamine and/or deferiprone) because of documented severe toxicity.
* Patients with a degree of iron overload which was not immediately life-threatening and who were ineligible for other trials with ICL670 could also be enrolled providing they had a well-documented, sound justification for alternative chelation therapy.
* Serum ferritin ≥ 8000 μg/L.
* Serum ferritin < 8000μg/L and LIC of ≥ 7 mg Fe/g dry weight.
* Patients for whom ≥ 8 blood transfusions per year were required in order to maintain the Hemoglobin level at > 9 g/dL.
* Female patients who have reached menarche and who were sexually active had to use double barrier contraception (oral plus barrier contraception), or had to have undergone total hysterectomy and/or ovariectomy, or tubal ligation.
* Written, voluntary informed consent.

Exclusion Criteria:

* Patients with transfusional iron overload who were not experiencing severe toxicities during therapy with other iron chelators (e.g. deferoxamine and/or deferiprone).
* Patients with non-transfusional hemosiderosis.
* Patients with severe liver failure as defined by a score of ≥ 10 points on the Child-Pugh scale.
* Patients with serum creatinine 1.5 times the upper limit of normal (ULN) at screening.
* Patients with a history of nephrotic syndrome.
* Patients with a diagnosis of clinically relevant cataract or a previous history of clinically relevant ocular toxicity related to iron chelation therapy.
* Patients with severe systemic diseases unrelated to iron overload and which would prevent them from undergoing treatment with ICL670.
* Patients with psychiatric or addictive disorders which prevent them from giving informed consent or undergoing treatment with ICL670.
* Pregnant or breast feeding patients.
* Patients treated with systemic investigational drugs within the past four weeks or topical investigational drugs within the past seven days.
* Any surgical or medical condition which might significantly alter the absorption or excretion of drugs as shown by evidence of any of the following:

  * History of inflammatory bowel disease
  * History of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection
  * History of pancreatic injury or pancreatitis; indication of impaired pancreatic function/injury as indicated by abnormal lipase or amylase
* Patients being considered by the investigator as potentially unreliable and/or not cooperative with regard to the protocol.
* History of drug or alcohol abuse within the 12 months prior to dosing.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2003-06; Primary Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety profile and to provide treatment with ICL670 for patients with or at risk of life-threatening complications due to transfusional iron overload who are unable to tolerate other iron chelators because of documented severe toxicity. | 0 - 163 weeks

SECONDARY OUTCOMES:
To estimate the absolute and relative change of liver iron concentration (LIC), to be measured using appropriate methodology available at individual centers. | Yearly
To evaluate the role of serum ferritin, serum iron, transferrin and transferrin saturation in monitoring iron burden in these patients. | Quarterly
To evaluate the relationship between changes in LIC and serum ferritin, transferring saturation and serum iron. | Yearly

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (18):
- United States (8):
  - Children's Hospital and Research Center - Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Children's Hospital Boston, Boston, Massachusetts
  - Queens Hospital Center, Jamaica, New York
  - New York Presbyterian Hospital/Weill Medical College of Cornell University, New York, New York
  - New York Methodist Hospital, New York, New York
  - Cincinnatti Children's Hospital Medical center, Cincinnatti, Ohio
  - Novartis Investigative Site, Houston, Texas
- Novartis investigative Site, Athens, Greece
- Italy (9):
  - Novartis Investigative Site, Ancona
  - Novartis Investigative Site, Brindisi
  - Novartis Investigative Site, Cagliari
  - Novartis Investigative Site, Cosenza
  - Novartis Investigative Site, Florence
  - Novartis Investigative Site, Milan
  - Novartis Investigative Site, Modena
  - Novartis Investigative Site, Napoli
  - Novartis Investigative Site, Torino

REFERENCES:
- See also: Related Info — http://www.novartisclinicaltrials.com/